CLINICAL TRIAL: NCT00584142
Title: Effects of MBSR in Early Stage Breast Cancer Recovery
Brief Title: Mindfulness-based Stress Reduction in Breast Cancer Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Cecile A. Lengacher RN PhD, University of South Florida, College of Nursing
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: R21CA109168 (NIH); R21CA109168 (NIH)
Record Dates: First submitted 2007-12-21; First posted 2008-01-02 (Estimated); Last update posted 2012-06-18 (Estimated); Status verified 2007-12

CONDITIONS: Breast Cancer
Keywords: breast cancer; survivors
MeSH Terms: conditions — Breast Neoplasms | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Behavioral: Mindfulness-Based Stress Reduction
- 2 (No Intervention)

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction — MBSR is a clinical program that provides systematic training to promote stress reduction by self-regulating arousal to stress. The goal of training is to teach participants to become more aware of their thoughts and feelings, and through meditation practice, to have the ability to step back from thoughts and feelings during stressful situations that contribute to increased emotional distress. The intervention incorporates simple yoga, sitting meditation, body scan, and walking meditation in a 6-week program.
  Other Names: MBSR
  Arms: 1

SUMMARY:
The purpose of this study was two-fold: (i) to assess whether MBSR favorably influences psychological status, quality of life, stress hormones, and immune status in breast cancer survivors; and (ii) to explore possible mechanisms by which MBSR may favorably influence these outcomes, in particular, through reduction in fear of breast cancer recurrence and associated perceived stress. Both objectives were studied at the critical transition time immediately following completion of surgical, radiation and/or chemotherapy therapy for breast cancer.

DETAILED DESCRIPTION:
Breast cancer is the most common cancer among women in the U.S. - about 1 in 8 women will develop the disease in their lifetime. Although tremendous strides have been made in its treatment, more than 40,000 deaths will be attributed to the disease in 2005 alone. These sobering and well-recognized risks are a major source of distress among women free from the disease, and among those who have completed treatment for new onset disease. Regarding the latter, clinical interventions are virtually absent during the highly stressful transitional period in coming off treatment to becoming a breast cancer survivor, and no studies have tested interventions to reduce distress, particularly fear of recurrence, and improve quality of life during this time. Therefore, we proposed to conduct a two-armed randomized wait-list controlled study on use of a mindfulness-based stress reduction (MBSR) intervention among 100 female breast cancer patients (stages 0-III) who have recently completed treatment with surgery, radiation and/or chemotherapy. Specifically, we investigated: (i) whether MBSR favorably influences psychological status, quality of life, stress hormones, and immune status; and (ii) possible mechanisms by which MBSR may work, in particular, through a reduction in fear of breast cancer recurrence. Both objectives were studied at the critical transition time following completion of surgical and adjuvant therapies (end of treatment to 18 months thereafter) for breast cancer. The MBSR intervention included 6 weeks of class sessions according to the curriculum established by Kabat Zinn and Santorelli. Analysis of covariance models are being used to assess whether change in the above-defined outcomes varies by random assignment (MBSR or wait-list), per the intention-to-treat principle. Moreover, change (reduction) in fear of recurrence attributed to MBSR is being investigated as a mediator. If this R21 exploratory study shows that MBSR improves patient proximal outcomes following completion of breast cancer treatment, the science will be mature enough for future large-scale evaluation of MBSR as a potential therapy to reduce long-term morbidity and mortality in breast cancer patient populations.

ELIGIBILITY:
Inclusion Criteria:

* 21 years old or older
* Diagnosed with Stage 0, I, II, or III breast cancer
* Undergone lumpectomy and completed adjuvant radiation and/or chemotherapy (end of treatment to 18 months post-treatment)
* Ability to read and speak English at the 8th grade level to respond to the survey questions

Exclusion Criteria:

* Advanced stage (IV) breast cancer
* History of mastectomy
* Current psychiatric diagnosis
* Recurrent treatment for prior breast cancer

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2006-03; Primary Completion 2012-02 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
To assess whether MBSR favorably influences psychological status (anxiety, perceived stress, depression), quality of life, and immune status (among post-treatment breast cancer survivors) | 6 weeks

SECONDARY OUTCOMES:
To explore possible mechanisms by which MBSR may favorably influence psychological status, quality of life, and/or immune status (in other words, "how" MBSR may work) (among post-treatment breast cancer survivors) | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Cecile A Lengacher, RN PhD, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida, Tampa, Florida, United States

REFERENCES:
- [Derived] Lengacher CA, Johnson-Mallard V, Post-White J, Moscoso MS, Jacobsen PB, Klein TW, Widen RH, Fitzgerald SG, Shelton MM, Barta M, Goodman M, Cox CE, Kip KE. Randomized controlled trial of mindfulness-based stress reduction (MBSR) for survivors of breast cancer. Psychooncology. 2009 Dec;18(12):1261-72. doi: 10.1002/pon.1529. PMID 19235193